CLINICAL TRIAL: NCT05096559
Title: The Evaluation of Sublingual Microcirculation To Guide Fluid Resuscitation In Patients With Burn: Prospective Observational Study
Brief Title: Evaluation of Sublingual Microcirculation in Burn During Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shymaa Fathy, Lecturer of anesthesia and SICU, Cairo University
Other Study IDs: N-111-2017
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Burn Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Microcirculation cytocam — Visualization of tongue microcirculation

SUMMARY:
The adequacy of fluid resuscitation will be monitored in burn patients using microcirculation.

Microcirculation camera will be placed on the base of the tongue and at different four quadrants. • Microcirculation parameters at baseline and after 8h , 16h and 24h of fluid resuscitation will be recorded. Fluid resuscitation with lactated ringer according to Parkland formula (4 ml/kg/%TBSA) 50% given during the first 8 hours, with the remainder given during the following 16 hours, will be initiated to maintain a urinary output of 0.5ml/kg/hr.Norepinephrine infusion will be started in case of circulatory failure at a rate of 0.02mic/kg/min to maintain MAP of 65-70mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Burn >20% TBSA
* Patients with burn admitted within the 1st 6 hours

Exclusion Criteria:

* Age < 18 years old.
* Pregnant patients.
* Patients with severe renal insufficiency.
* Patients shocked due to other causes as sepsis, hypovolaemia or cardiogenic shock
* Patients with airway edema that preclude the measurement of sublingual microcirculation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with burns greater than 20% TBSA admitted to ICU within the 1st 6 hours post-burn
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
• Lactate level | 24 hours
  mmol/L

SECONDARY OUTCOMES:
total vessel density | 24 hours
  mm/mm2

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No